CLINICAL TRIAL: NCT06168071
Title: Safety, Tolerability and Neurophysiological Response of Transauricular Vagus Nerve Stimulation in Children Without Brain Injury
Brief Title: Transauricular Vagus Nerve Stimulation in Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202307034
Record Dates: First submitted 2023-11-28; First posted 2023-12-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hypoxia-Ischemia, Brain
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- taVNS with EEG in healthy children (Experimental): The investigators will enroll 10 children between 7-18 years of age who are admitted to the hospital for EEG monitoring for spell characterization to receive one session of 30 minutes of taVNS. The investigators will titrate taVNS to below perceptual threshold of stimulation and objectively assess tolerability. The following parameters will be used for taVNS: frequency 25 Hz, pulse width 250 µs, and varying intensities from 0.5 milliampere (mA) to 2 mA. Intensity will be titrated to be a level below perceptual threshold in a patient. The participant will have continuous cardiorespiratory monitoring via pulse oximetry and blood pressure every 5 minutes. EEG data will be compared before, during and after taVNS.
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — Recently, implantable VNS received FDA approval for augmenting motor recovery from ischemic stroke-induced hemiplegia when used during standard physical and occupational therapy sessions. VNS is FDA-approved for epilepsy therapy in children and is used for generalized refractory epilepsy. VNS may be achieved through an implantable stimulator on the left vagus nerve in the carotid sheath, or transcutaneously through the auricular branch of the vagus nerve (taVNS). All participants will be fitted with the device by attaching adhesive contacts to the left ear. Stimulation sessions will occur once for 30 minutes. The investigators will obtain baseline measure, tolerability questionnaires, vital signs, and EEG data.

SUMMARY:
The goal of this clinical trial is to learn about brain waves during transauricular vagus nerve stimulation (taVNS) in healthy children.

The main questions it aims to answer are:

* What is the safety, tolerability, and physiological response of taVNS in children?
* Does the electroencephalogram (EEG) change during taVNS?

Participants will

* undergo a brief titration session where taVNS will be titrated to below perceptual threshold
* receive one session of 30 minutes of taVNS
* undergo clinical EEG monitoring during taVNS
* Continuous cardiorespiratory monitoring via pulse oximetry and blood pressure every 5 minutes
* Answer tolerability questions before, during and after 30 minute taVNS session

ELIGIBILITY:
Inclusion Criteria:

* Admitted for clinical EEG for spell characterization at investigator's institution

Exclusion Criteria:

* known history of brain injury
* known history of bradycardia
* congenital heart disease
* pregnant
* pacemaker or wearable defibrillator
* undergoing active cancer treatment

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety: Heart rate | Baseline and continuously for 30 minutes during study visit. It will be recorded and assessed every 5 minutes during 30 minute study visit.
  Determined by continuous pulse oximeter. If heart rate drops below 60 beats per minute (bpm) in children younger than 9 years and below 50 bpm in children older than 9 years for more than 30 seconds, the stimulation will be stopped.
Safety: Oxygen saturation | Baseline and continuously for 30 minutes during study visit. It will be recorded and assessed every 5 minutes during 30 minute study visit.
  Determined by continuous pulse oximeter. If oxygen saturation drops below 92% for more than 30 seconds, stimulation will stop.
Tolerability: Face, Legs, Activity, Cry, Consolability (FLACC) | Baseline prior to stimulation, 15 minutes into the stimulation and immediately following the 30 minute stimulation.
  Observation pain assessment before, during and after stimulation. FLACC scale is a 0-10 pain scale with 10 being severe pain and 0 being no pain.
Tolerability: Tolerance Questionnaire | Baseline prior to stimulation, 15 minutes into the stimulation and immediately following the 30 minute stimulation.
  Qualitative survey of side effects, ranking of preference of taVNS activity and 6-point comfort scale (6 being severely uncomfortable). Completed before, during and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Smith, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT06168071/ICF_000.pdf